CLINICAL TRIAL: NCT05699538
Title: Fatigue and Fatigability in Veterans Following SARS-CoV-2 Infection
Brief Title: Fatigability in Long COVID-19
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F4371-P
Record Dates: First submitted 2023-01-24; First posted 2023-01-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Long COVID
Keywords: resistance exercise; fatigue; COVID-19; near infrared spectroscopy; strength
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimal-Dose Home-Based Resistance Exercise (Experimental): 8-week home-based resistance exercise performed one day per week.
  Interventions: Behavioral: Minimal-Dose Home-Based Resistance Exercise
- Standard of Care (No Intervention): Subjects will be asked to follow standard of care recommendations as prescribed by the physician.

INTERVENTIONS:
Behavioral: Minimal-Dose Home-Based Resistance Exercise — 8-week home-based resistance exercise performed one day per week.
  Arms: Minimal-Dose Home-Based Resistance Exercise

SUMMARY:
The overall goal of this project is to advance the understanding of underlying mechanisms impacting performance fatigability and perceived fatigability in Veterans with post-COVID-19 fatigue and explore the safety and feasibility of a home-based "minimal-dose" resistance exercise program in this population. The central hypothesis is that declines in force capacity, skeletal muscle oxygen extraction, and affective responses to physical activity offer potential mechanisms through which fatigability is increased in Veterans with post-COVID-19 fatigue. Moreover, home-based resistance exercise delivered remotely may provide a safe and feasibility treatment option for targeting neuromuscular and neurobehavioral factors influencing fatigability severity in this population.

DETAILED DESCRIPTION:
The clinical case definition of post-COVID-19 condition (also referred to as Long COVID) as defined by the World Health Organization (WHO) includes individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms and that last for at least 2 months and cannot be explained by an alternative diagnosis. Fatigue represents one of the most frequently reported symptoms in individuals experiencing post-COVID-19 (i.e., post-COVID-19 fatigue; PCF).Fatigue is shown to persist for months after SARS-CoV-2 infection, negatively impacting activities of daily living. For the purposes of this SPiRE proposal, fatigue is operationally defined as a state characteristic encompassing a subjective lack of physical and/or mental energy that is perceived by the individual to interfere with usual or desired activities.

Increased fatigability is a possible complication following SARS-CoV-2 infection due to the presence of both neuromuscular and neurobiological consequences. Skeletal muscle alterations including reduced force capacity, fiber atrophy, mitochondria and metabolic dysfunction, and capillary impairments have been observed in patients following SARS-CoV-2 infection. Autopsy reports of patients who died after SARS-CoV-2 infection found evidence of skeletal muscle atrophy of type 2 fibers, necrotizing myopathy, and myositis. Similarly, using nerve conduction studies, patients with long-term COVID-19 were found to have signs of myopathy, even those who were not hospitalized. Evidence from cardiopulmonary exercise testing in patients diagnosed with COVID-19 has revealed impaired skeletal muscle oxygen extraction, as opposed to central limitations (i.e., cardiac output), as a determinant of exercise intolerance. In addition to neuromuscular complications, SARS-CoV-2 infection has also been shown to be associated with psychiatric sequelae. Collectively, these findings underscore neuromuscular as well as neurobiological consequences of SARS-CoV-2 as potential independent or co-occurring mechanisms by which increased fatigability occurs and persists.

Despite widespread calls for the importance of rehabilitation in individuals recovering from SARS-CoV-2 infection, little progress has been made regarding the potential benefits of physical exercise on fatigue and fatigability in this population. Moreover, concerns have been raised about the applicability of physical exercise in patients recovering from SARS-CoV-2 infection. For example, while the health and functional benefits of exercise are vast and widely known, in certain patient populations exertion is shown to exacerbate symptom severity. Some individuals with PCF may report experiencing worsening of symptoms after physical or mental exertion. Home-based exercise may offer an appealing option for those individuals concerned about attending community fitness facilities. Home-based exercise is shown to produced moderate effects on muscle strength and balance. Presently, the exact dosing of home-based exercise to elicit positive outcomes in fatigability is unknown. Minimal-dose resistance exercise has been proposed as a potential strategy for improving neuromuscular characteristics and physical function. Minimal-dose resistance exercise uses little to no equipment with exercises performed at lower workloads. The investigators aim to adapt the "minimal-dose" resistance exercise paradigm to a remote home-based resistance exercise program for Veterans with PCF to determine its implications for reducing fatigability and improving neuromuscular and neurobiological factors. Minimal-dose resistance exercise for the proposed application is defined as a single, weekly body-weight exercise session.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory patients (with or without a gait aid)
* 50 years of age or older
* with a confirmed diagnosis of COVID-19 by polymerase chain reaction (PCR) test, antibody test or clinical diagnosis
* the symptom of fatigue reported greater than 12-weeks post-infection (reporting fatigue: yes/no)
* receiving care at the DC VAMC
* the ability to speak and read English, and orientation to person, place, and time

  * the comparison group will include ambulatory patients (with or without a gait aid)
  * 50 years of age or older
  * with a confirmed diagnosis of COVID-19 by PCR test, antibody test or clinical diagnosis
  * without the symptom of fatigue reported greater than 12-weeks post-infection
  * receiving care at the DC VAMC
  * the ability to speak and read English, and orientation to person, place, and time

Exclusion Criteria:

* <50 years of age without a confirmed diagnosis of COVID-19 by PCR test
* antibody test or clinical diagnosis or with a confirmed diagnosis of COVID-19 of <12-weeks
* non-ambulatory individuals
* Veterans who do not use the DC VAMC as their main site for care
* body mass index 40 kg/m2
* diagnosis of psychiatric disorder(s)
* any medically uncontrolled cardiovascular
* musculoskeletal disease, or other conditions that, in the opinion of the principal investigator, could make participation in the study unsafe
* any orthopedic or joint pain which would prevent the participant from safely engaging in the study protocol
* additionally, individuals with plans to relocate from the DC metro area within one year will not be eligible for the intervention portion of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance fatigability | baseline and week 8
  Performance fatigability will be assessed as change in maximal voluntary isometric contraction (MVIC) torque of the dominant leg. Change in MVIC torque from the initial MVIC contraction to the last MVIC contraction will be used to determine the Performance Fatigability index.

SECONDARY OUTCOMES:
Rating of Perceived Fatigue (RPF) | baseline and week 8
  Perceived fatigability will be assessed using a rating of perceived fatigue (RPF) scale.
  0=no fatigue at all; 10=absolutely exhausted higher the value=more fatigue
Isometric and Isokinetic Knee Extensor Torque | baseline and week 8
  Unilateral peak isometric and isokinetic knee extension torque (60º/s and 180º/s) will be obtained across five continuous repetitions using a dynamometer in a seated position per manufacturer guidelines (Biodex System 4).
Skeletal muscle oxygen extraction | baseline and week 8
  Skeletal muscle oxygen extraction of the dominant vastus lateralis will be assessed non-invasively using near-infrared spectroscopy (NIRS) (Artinis, Portamon, The Netherlands).
Feeling Scale | baseline and week 8
  Change's in affect during knee extensor performance fatigability testing will be assessed using the Feeling Scale. The Feeling Scale is an 11-point, single item, bipolar rating scale ranging from +5 to -5.
Fatigue Severity Scale (FSS) | baseline and week 8
  9-item questionnaire assessing how fatigue interferes with certain activities and rates its severity according to a self-report scale. Items are scored on a 7-point scale with 1=strongly disagree and 7=strongly agree. higher the value=more impact fatigue has
Short Physical Performance Battery (SPPB) | baseline and week 8
  SPPB will assess customary gait speed, side-by-side stand, semi-tandem stand, tandem stand, and 5-STS.
30-second sit-to-stand | baseline and week 8
  subjects will be asked to perform as many sit-to-stand repetitions in 30 seconds.
Six Minute Walk Test (6MWT) | baseline and week 8
  Subjects will be asked to walk as far as possible in 6 minutes.
Motor Unit Firing Rate | baseline and week 8
  motor unit shape and firing behavior of the dominant leg vastus lateralis will be extracted using surface electromyographic signals (sEMG) and specialized software (Trigno NeuroMap System, Delsys Inc., Natick, MA, USA).
Muscle Activation | baseline and week 8
  interpolated twitch technique will be applied to the femoral nerve using a constant-current, variable high-voltage stimulator (DS7R, Digitimer, Hertforshire, UK) to quantify muscle activation of the vastus lateralis.
peak VO2 | baseline and week 8
  Peak VO2 will be assessed from cardiopulmonary exercise testing using the Modified Bruce Protocol.
Health-related quality of life (SF-36) | baseline and week 8
  The 36-item short-form (SF-36) is a multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
Pittsburgh Fatigability Scale | baseline and week 8
  26-item scale chosen from four activity categories; social, sedentary, lifestyle or light-intensity, and moderate-to-high-intensity.
Short-form Depression, Anxiety, and Stress Scale (DASS-21) | baseline and week 8
  The DASS is designed to measure the negative emotional states of depression, anxiety, and stress.
Physical Activity Level | baseline and week 8
  Physical activity levels will be monitored objectively using ActiGraph activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Jared M. Gollie, PhD, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT05699538/ICF_000.pdf